CLINICAL TRIAL: NCT03202966
Title: Early Intervention Therapy for Children With Delayed Development: Enabling Access in India's Rural Communities
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Amar Seva Sangam (Other)
Collaborators: Grand Challenges Canada (Other); University of Toronto (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 0819-05
Record Dates: First submitted 2017-06-25; First posted 2017-06-29 (Actual); Last update posted 2020-04-28 (Actual); Status verified 2020-04

CONDITIONS: Developmental Delay
MeSH Terms: conditions — Learning Disabilities | interventions — Rehabilitation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): For each child with a developmental delay enrolled in the early intervention program, individualized rehabilitation therapy will be provided by a rehabilitation professional with a focus on the one or more domains where delays were identified (i.e. speech, motor, cognition). The intervention will be delivered either as home based rehabilitation or as centre based care. Each child will receive a minimum of one therapy session per week by the CRW and a monthly therapist visit for home based care. In center based care daily therapy will be available by either a CRW or specialist.
  Interventions: Other: Rehabilitation therapy

INTERVENTIONS:
Other: Rehabilitation therapy — Rehabilitation therapy will be provided by a trained community rehabilitation worker (CRW) and specialist (i.e., physical therapist, occupational therapist, special educator and/or speech therapist) with a focus on the one or more domains where delays are identified (i.e. speech, motor, cognition). Therapy will be tailored based on the needs of the individual child and will follow current evidence-based practice.

SUMMARY:
This study is a cohort longitudinal design, also known as within subject repeated measures' design to measure the impact of an early identification and intervention program being implemented by Amar Seva Sangam (ASSA), an Indian non-government organization in South India. The primary objective of the Early Intervention (EI) Village-Based Rehabilitation (VBR) program is to increase access to early identification and early intervention therapy to enhance physical, cognitive, language, social and emotional development of children with developmental delays. The primary outcome will be the creation of developmental trajectory of girls and boys with developmental delay who are receiving village based early intervention therapy in rural India, aged 0 - 6 years based on the Gross Motor Function Measure - GMFM (children with cerebral palsy only), Functional Independence Measure - wee-FIM, Functional Assessment Checklist for Programming - FACP, Communication Developmental Eclectic Approach to Language Learning - CDDC and Canadian Occupational Performance Measure - COPM. Secondary outcomes will be the effect of therapy compliance rates on development in girls and boys with developmental delay, the effect of therapeutic approach on development in girls and boys with developmental delay, improved enrolment in school for children with developmental delays from age 3 to 6; and, improved parent/caregiver knowledge, attitude, behavior and confidence in caring for their child with developmental delay.

DETAILED DESCRIPTION:
This study is a cohort longitudinal design, also known as within subject repeated measures' design to measure the impact of an early identification and intervention program being implemented by Amar Seva Sangam (ASSA), an Indian non-government organization in South India. The primary objective of the Early Intervention (EI) Village-Based Rehabilitation (VBR) program is to increase access to early identification and early intervention therapy to enhance physical, cognitive, language, social and emotional development of children with developmental delays. The primary outcome will be the creation of developmental trajectory of girls and boys with developmental delay who are receiving village based early intervention therapy in rural India, aged 0 - 6 years based on the Gross Motor Function Measure - GMFM (children with cerebral palsy only), Functional Independence Measure - wee-FIM, Functional Assessment Checklist for Programming - FACP, Communication Developmental Eclectic Approach to Language Learning - CDDC and Canadian Occupational Performance Measure - COPM. Secondary outcomes will be the effect of therapy compliance rates on development in girls and boys with developmental delay, the effect of therapeutic approach on development in girls and boys with developmental delay, improved enrolment in school for children with developmental delays from age 3 to 6; and, improved parent/caregiver knowledge, attitude, behavior and confidence in caring for their child with developmental delay.

For each child with a developmental delay who is enrolled in the early intervention program, a detailed care plan will be developed by the rehabilitation professional(s) who will provide the care based on the specific needs of the child. A trained community rehabilitation worker (CRW) will implement the care plan with a focus on the one or more domains where delays were identified (i.e. speech, motor, cognition). The intervention will be delivered either within the child's home (home based rehabilitation) or at an local Early Intervention Parent Participation Centre (EI PPCs) (centre based care). Each child will receive a minimum of one therapy session per week by the CRW and a monthly therapist visit (i.e., physical therapist, occupational therapist, special educator and/or speech therapist) for home based care. In center based care daily therapy will be available by either a CRW or specialist. In addition, monthly team meetings will be held by the specialists and CRWs to monitor progress and modify or adapt therapy plans as needed. Therapy will be tailored based on the needs of the individual child and will follow current evidence-based practice. The investigators will do evaluations using the standardized scales noted above (GMFM, WEE FIM, COPM, FACP and COM DEALL) every 6 months to monitor the progress of the child.

ELIGIBILITY:
Inclusion Criteria:

* Boys and girls
* Newborn to age 6
* Identified with developmental delay based on the Trivandrum screening tool
* Diagnosed as definitive delayed development by a team of rehabilitation specialists (i.e. physical therapist, occupational therapist, speech therapist, special educator)
* Receiving either home-based or center-based care in the ASSA Village-Based Early Intervention Program
* Live in one of the following 7 blocks in the District of Tirunelveli: Alangulam Block; Kadayanallur Block; Keelapavoor Block; Shenkottai Block; Tenkasi Block; Sankarankoil Block; and, Vasudevanallur Block

Exclusion Criteria:

* None

Max Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1050 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2019-07-30 (Actual); Study Completion 2019-07-30 (Actual)

PRIMARY OUTCOMES:
Developmental Score Trajectory as Assessed by the Canadian Occupational Performance Measure (COPM) | From date of recruitment up to 2 years
  The Canadian Occupational Performance Measure (COPM) is a standardized client-centred outcome measure. Using a semi-structured interview format, the participant would asked to identify individual goals for occupational performance, related to self-care, productivity and leisure, that the participant has difficulty completing. Participants are asked to identify the 5 most important problems and for each problem/goal they are asked to rate both their performance and satisfaction on a scale of 1 to 10 (1= poor performance, low satisfaction; 10 = good performance, high satisfaction). Total scores are calculated by adding the performance or satisfaction scores for all problems and dividing by the number of problems. The average scores (1 to 10) for each scale of the COPM (performance and satisfaction) are used for analysis and comparison between assessments.
Developmental Score Trajectory as Assessed by the Gross Motor Function Measure (GMFM-88) | From date of recruitment up to 2 years
  The Gross Motor Function Measure (GMFM-88) is a validated assessment designed specifically for participants with cerebral palsy to evaluate change and development of participant's gross motor function. This is an 88-item assessment with each item scored on a 4-point system (0=does not initiate; 1=initiates; 2=partially completes; 3=completes; and NT=not tested). The GMFM-88 is a validated functional outcome measure, with demonstrated reliability and responsiveness that can be used to evaluate meaningful change in gross motor function over time.
Developmental Score Trajectory as Assessed by the Functional Independence Measure for Children (wee-FIM) | From date of recruitment up to 2 years
  The Functional Independence Measure for Children (wee-FIM) is a standardized and internationally validated assessment that evaluates participant's performance in self-care, sphincter control, transfers, location, communication and social cognition. The wee-FIM is an 18-item measure using a 7-level ordinal scale (1=total assist and 7=complete independence). It is organized into 2 subscales - motor and cognitive. It has been validated in a variety of settings, including in developing countries and has been demonstrated to have transcultural applicability. The wee-FIM has an acceptable responsiveness to demonstrate change over time.
Developmental Score Trajectory as Assessed by the Communication DEALL Development Checklist (CDDC) | From date of recruitment up to 2 years
  The Communication DEALL (Developmental Eclectic Approach to Language Learning) Developmental Checklist (CDDC) will be used for speech assessment. The CDDC evaluates skills in eight developmental domains including: gross motor, fine motor, activities of daily living, receptive language, expressive language, cognitive skills, social skills and emotional skills. Only the domains for expressive language and receptive language will be used for the assessments. A 5-point scale is used to measure skill development (0= not acquired; 1 acquired but lost; 2 acquired but inconsistently present; 3= acquired and consistently present but only in specific situations; 4=acquired and consistently present across all situations). Within each domain questions are divided into 12 subgroups based on 6-month age groups (i.e., 0-6 months, 6-12 months etc.). This instrument has been validated in urban children, age 0-6 years, in India and has strong inter rater reliability.
Developmental Score Trajectory as Assessed by the Functional Assessment Checklist Programming (FACP) | From date of recruitment up to 2 years
  The Functional Assessment Checklist for Programming (FACP) is a standardized measure that evaluates a participant's performance in 4 domains: occupational, academic, social, and personal skills. This instrument was developed and validated in India for use in special education. A checklist is used to evaluate the performance or achievement of the participant in each task. Performance is measured on a 5-point scale (0 to 5), where 0 means totally unable and 5 means totally able. The usual evaluation is comprised of 120 items, but the investigators will use an 88 item version. A total percentage score is generated for each participant's overall performance.

SECONDARY OUTCOMES:
Treatment Compliance as Assessed by Therapy Sessions Achieved by Therapy Assessments Planned | From date of recruitment up to 2 years
  The treatment compliance measure will be calculated as a proportion based on the number of therapy sessions achieved by each participant by the number of therapy sessions planned for that participant.
School Enrolment of Participants as Assessed by Enrolment Status | From date of recruitment up to 2 years
  School enrolment will be measured as a proportion of the participants who are enrolled in school by school type (preschool, primary school, special needs school).
Parent/Caregiver Change as Assessed by the Tirunelveli Early Intervention Caregiver Assessment Tool | From date of recruitment up to 2 years
  The Tirunelveli Early Intervention Caregiver Assessment Tool will be used with the primary caregivers of the participants (i.e. the person who is most involved in the day-to-day care of the child with developmental delay). This instrument will measure 1) family empowerment using the 12-item family sub scale of the Family Empowerment Scale (FES); 2) caregiver burden using the Modified Caregiver Strain Index (MCSI); and, 3) interactions with the participant based on a newly constructed 10-item questionnaire.

CONTACTS AND LOCATIONS:
Locations (2):
- India (2):
  - Ayikudy, Tamil Nadu
  - Amar Seva Sangam, Ayikudy

IPD SHARING:
Plan to Share IPD: No